CLINICAL TRIAL: NCT00004492
Title: Phase I/II Randomized Study of Hydroxyurea With or Without Clotrimazole in Patients With Sickle Cell Anemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of North Carolina (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 199/14273; UNCCH-FDR001531
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2001-01

CONDITIONS: Sickle Cell Anemia
Keywords: genetic diseases and dysmorphic syndromes; hematologic disorders; rare disease; sickle cell anemia
MeSH Terms: conditions — Anemia, Sickle Cell; Genetic Diseases, Inborn; Hematologic Diseases; Rare Diseases | interventions — Clotrimazole; Hydroxyurea

INTERVENTIONS:
Drug: clotrimazole
Drug: hydroxyurea

SUMMARY:
OBJECTIVES:

I. Compare the efficacy of hydroxyurea with or without clotrimazole in terms of limiting the severity of anemia and the rate of hemolysis in patients with sickle cell anemia.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized study. Patients are randomized to one of two treatment arms.

Arm I: Patients receive oral hydroxyurea and oral clotrimazole daily for 12 months.

Arm II: Patients receive oral hydroxyurea daily for 12 months. Patients are followed at 6 weeks.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Diagnosis of sickle cell anemia confirmed by hemoglobin electrophoresis

Received hydroxyurea for at least 6 months On a stable dose for at least 3 months Tolerating dose of at least 5 mg/kg/day

--Prior/Concurrent Therapy--

Chemotherapy:

* No other concurrent antisickling agent

Other: No concurrent drug that may interact with or influence the metabolism of hydroxyurea or clotrimazole

--Patient Characteristics--

Hematopoietic: WBC at least 4000/mm3 Platelet count at least 150,000/mm3 Hemoglobin less than 11 g/dL

Hepatic: AST/ALT no greater than 100 units/L

Renal: Creatinine no greater than 1.5 mg/dL

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No prior adverse reaction to hydroxyurea or clotrimazole
* No recent or progressive neurologic dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 1999-10; Study Completion 2001-09

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Paul Orringer, Study Chair — University of North Carolina
Locations (1):
- University of North Carolina School of Medicine, Chapel Hill, North Carolina, United States